CLINICAL TRIAL: NCT02085655
Title: PA-Gemox Regimen Followed by Thalidomide Versus AspaMetDex Regimen in NKTCL Patients：a Randomized, Open-label, Phase 3 Study
Brief Title: PEG-ASP+Gemox Regimen and Thalidomide for NK/T Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huiqiang Huang (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor-Investigator, Huiqiang Huang, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NKT-SYSUCC-2013
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Extranodal NK-T-Cell Lymphoma, Nasal and Nasal-Type
Keywords: Extranodal NK/T-cell lymphoma; PA-Gemox regimen; thalidomide
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — pegaspargase; Gemcitabine; Oxaliplatin; Methotrexate; Dexamethasone; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEG-ASP+Gemox regimen group (Experimental): PEG-ASP 2000U/m2 im d1 Gemcitabine 800mg/m2 ivdrip 30min d1，8 Oxaliplatin 100mg/m2 ivdrip d1 Thalidomide 150-200mg po qn d8-21
  Interventions: Drug: pegaspargase; Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Thalidomide
- AspaMetDex regimen group (Active Comparator): Pegaspargase 2000U/m2 im， d1 methotrexate 3000m g/m2 civ 6-hour，d1, Calcium folinate 30mg iv q6h x6 Dexamethasone 40 mg ivdrip QD
  Interventions: Drug: pegaspargase; Drug: Methotrexate; Drug: Dexamethasone

INTERVENTIONS:
Drug: pegaspargase — pegaspargase: 2000U/m2 im on day 1 of each 21 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Oncaspar
Drug: Gemcitabine — 1000mg/m2, ivd on day 1 and 8 of each 21 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Gemzar
  Arms: PEG-ASP+Gemox regimen group
Drug: Oxaliplatin — 100mg/m2 ivd on day 1 of each 21 day cycle. Number of Cycles: until progression or unacceptable toxicity develops
  Other Names: Eloxatin
  Arms: PEG-ASP+Gemox regimen group
Drug: Methotrexate — 3000m g/m2 civ 6-hour on day 1 of each 21 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Arms: AspaMetDex regimen group
Drug: Dexamethasone — 40mg ivd on day 1 of each 21 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Arms: AspaMetDex regimen group
Drug: Thalidomide — 100-200mg, PO, after chemotherapy
  Arms: PEG-ASP+Gemox regimen group

SUMMARY:
Extranodal natural killer/T-cell lymphoma (ENKTL) is an aggressive form of non-Hodgkin's lymphoma and shows extremely poor survival. This prospective pilot study to evaluate the efficacy and safety of long-acting aspargase (pegylated aspargase, PEG-ASP) combined with gemcitabine and oxaliplatin (PASP -Gemox) treatment in this population.

DETAILED DESCRIPTION:
Eligibility criteria The eligibility criteria were pathologically confirmed, previously untreated or refractory/relapsed ENKTL as defined by the World Health Organization classification; age≥18 years; Eastern Cooperative Oncology Group (ECOG) performance status of 0-2; at least one measurable lesion; adequate haematologic function (haemoglobin > 9.0 g/l, absolute neutrophil count > 1500/ml, platelets > 75,000/l), hepatic function (total serum bilirubin ≤ 1.5 times the upper limit of normal, alanine aminotransferase and aspartate aminotransferase ≤ 2.5 times the upper limit of normal), renal function (serum creatinine ≤ 1.5 mg/dl, creatinine clearance ≥ 50 ml/min); normal coagulation function and electrocardiogram results. Prior chemotherapy and radiotherapy should have been completed >4 weeks earlier, willingness to provide written informed consent. Stage was defined according to the Ann Arbor system. The Sun Yat-Sen University Cancer Centre Research Ethics Board approved this study before subjects were enrolled.

Treatment PA-Gemox dosages were as follows: days 1 and 8, 30-min intravenous infusion of 1000 mg/m2 gemcitabine; day 1, 2-h intravenous infusion of 130 mg/m2 oxaliplatin; day 1, deep intramuscular injection of 2500 U/m2 PEG-ASP at two different sites. The regimen was repeated every 3 weeks for a maximum of six cycles. Stage IE/IIE patients underwent four cycles induction chemotherapy, followed by involved-field radiotherapy after got CR, PR or SD. Three-dimensional conformal radiotherapy was done by linear accelerator at 2.0 grays (Gy) per daily fraction with 5-6 weeks. The involved- field radiation (IFRT) dose was 50-56 Gy. Refractory/relapsed patients underwent at least two cycles treatments unless there was disease progression or unacceptable side effects, or withdrawal of patient consent. Autologous haematopoietic stem cell transplantation (AHSCT) was recommended after they achieved CR.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically confirmed, previously untreated or refractory/relapsed ENKTL as defined by the World Health Organization classification;
2. age≥18 years;
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
4. at least one measurable lesion;
5. adequate haematologic function (haemoglobin > 9.0 g/l, absolute neutrophil count > 1500/ml, platelets > 75,000/l),
6. adequate hepatic function (total serum bilirubin ≤ 1.5 times the upper limit of normal, alanine aminotransferase and aspartate aminotransferase ≤ 2.5 times the upper limit of normal),
7. adequate renal function (serum creatinine ≤ 1.5 mg/dl, creatinine clearance ≥ 50 ml/min);
8. normal coagulation function and electrocardiogram results.
9. Prior chemotherapy and radiotherapy should have been completed >4 weeks earlier,
10. willingness to provide written informed consent.

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2013-04-25 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy Outcome Measure | up to 24 months
  Study group increase 15% 2-year PFS

SECONDARY OUTCOMES:
Safety/Adverse Event Outcome Measure | Up to 36 months
  Number of Participants with Serious and Non-Serious Adverse Events

OTHER OUTCOMES:
Efficacy Outcome Measure | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: HuiQiang Huang, Study Chair — Sun Yat-sen University
Locations (1):
- Department of Medical Oncology, Sun Yat-sen University Cancer Center,, Guangzhou, Guangdong, China